CLINICAL TRIAL: NCT05644873
Title: The Effect of Intravenous Magnesium Sulfate Use on Intraoperative Remifentanil Consumption and Postoperative Pain in Abdominal Hysterectomy Cases
Brief Title: Intravenous Administration of Magnesium Sulfate in Hysterectomy Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ITamdogan
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Abdominal Hysterectomy; General Anesthesia; Magnesium Sulfate
Keywords: postoperative pain; intravenous magnesium sulfate
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into two groups according to a 1:1 randomization ratio using opaque sealed envelopes before surgery. Study randomization was performed using computer generated randomization codes by SPSS v23.0 (IBM, New York, USA). Each patient was asked to choose an envelope and the patients were assigned to the study according to the group specified in the envelope. The drugs to be used were prepared 30 minutes before the surgery by the nurse who did not participate in the study in the drug preparation room. Everyone involved in this study, including patients, researchers, the anesthesiologist responsible for anesthesia management, and the surgeon, remained blind to group distribution during the study.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium sulfate (Active Comparator): Before induction, a bolus of 20 mg/kg magnesium sulfate in 100 mL saline was administered for 15 minutes, followed by a continuous infusion of 20 mg/kg/hour until the skin was closed.
  Interventions: Drug: magnesium sulfate group
- Placebo (Active Comparator): The control group received only 100 ml of saline 15 minutes before induction.
  Interventions: Drug: control group saline

INTERVENTIONS:
Drug: magnesium sulfate group — Anesthesia induction was provided with propofol (2mg/kg), fentanyl (2mcg/kg). Intubation was performed after administration of 0.6 mg/kg rocuronium with an appropriate endotracheal tube. Anesthesia was maintained using AIR/O2 (50%/50%), 1 minimum alveolar concentration (MAC) sevoflurane, 0.1-0.25 mcg/kg/min remifentanil infusion. The target BIS value was kept between 40 and 50. Systolic blood pressure (SBP) <90mmHg or <20% of baseline was considered hypotension; remifentanil infusion was reduced. If no response was obtained, 5-10 mg of IV ephedrine was administered. HR < 45 beats/min was evaluated as bradycardia; IV atropine 0.5 mg was planned The magnesium group received a bolus of 20 mg/kg of magnesium sulfate in 100 mL of saline for 15 minutes prior to induction, followed by a continuous infusion of 20 mg/kg/hr until skin closure.
  Other Names: magnesium sulfate
  Arms: Magnesium sulfate
Drug: control group saline — Anesthesia induction was provided with propofol (2mg/kg), fentanyl (2mcg/kg). Intubation was performed after administration of 0.6 mg/kg rocuronium with an appropriate endotracheal tube. Anesthesia was maintained using AIR/O2 (50%/50%), 1 minimum alveolar concentration (MAC) sevoflurane, 0.1-0.25 mcg/kg/min remifentanil infusion. The target BIS value was kept between 40 and 50. Systolic blood pressure (SBP) <90mmHg or <20% of baseline was considered hypotension; remifentanil infusion was reduced. If no response was obtained, 5-10 mg of IV ephedrine was administered. HR < 45 beats/min was evaluated as bradycardia; IV atropine 0.5 mg was planned The same volume of isotonic saline for the control group was administered as indicated in the magnesium group.
  Other Names: saline
  Arms: Placebo

SUMMARY:
In our study, it was aimed to show the contribution of intraoperative intravenous magnesium sulfate administration to peroperative opioid consumption and postoperative analgesia.

DETAILED DESCRIPTION:
Postsurgical pain is one of the most important issues that could impress on postoperative peace and comfort. Abdominal hysterectomy associated with intense inflammatory response, resulting in moderate to severe postoperative pain perception The major goal in postoperative pain management is to minimize the dose of medications and lessen side effects, while still providing adequate analgesia. Postoperative pain relief leads to earlier mobilization, shortened hospital staying, reduced hospital costs, and increased patient satisfaction Narcotics are the most common analgesics which are used after the surgeries. But anesthetists are always looking for replaceable methods with fewer side effects and cost . It seems adjuvant analgesics are those desirable replacements. Nowadays there have been many debates on the role of adjuvant analgesics on postoperative pain relief. One way to use adjuvant analgesics is preventive method Preventive analgesia is a method initiated before anesthetic procedure in order to reduce the physiological consequences of nociceptive stimulation and medical adverse effects and has been defined as an antinociceptive treatment that prevents establishment of altered central processing ofafferent input from injuries. One of the intravenous adjuvant that has been shown potential in preventive analgesia is magnesium sulfate that could be administered with multiple routes or methods Mg has been used for many years in anesthesia and cardiology as an anticonvulsant or antiarrhythmic drug. The mechanism of the analgesic effect of Mg is not clear but inter- ference with calcium channels and N-methyl-D-aspartate (NMDA) receptor seem to play an important role. It seems that analgesic mechanism of NMDA-antagonists is made by preventing nociceptive central sensitization. Another suggesting mechanism is the role of it on reduction of catecholamine release with sympathetic stimulation, thereby decreasing peripheral nociception or the stress response to the surgery. Data illustrate that the NMDA receptor antagonists "like Mg sulfate" have an effect on pain threshold and could prevent pain perception even with low doses (preventive doses) In our study, investigators aimed to determine the contribution of magnesium sulfate to postoperative analgesia in abdominal hysterectomy by considering its mechanism of action.

The patients were divided into two groups as magnesium sulfate administered and non-administered The magnesium group received a bolus of 20 mg/kg of magnesium sulfate in 100 mL of saline for 15 minutes before induction, followed by a continuous infusion of 20 mg/kg/hr until the skin was closed. The same volume of isotonic saline for the control group was administered as indicated in the magnesium group.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing abdominal hysterectomy
* Between the ages of 20-70,
* ASA I- II

Exclusion Criteria:

* Presence of hepatic and renal dysfunction,
* Presence of cardiac arrhythmia or other cardiac comorbidity,
* Neurological and psychiatric disorder,
* Chronic use of calcium and beta blockers,
* Drug or alcohol abuse,
* Pregnancy and lactation status,
* Patients with a history of allergy to any drug included in the study protocol

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome of this study was total opioid consumption in the first 24 hours postoperatively | Postoperative Day 1
  IV patient-controlled analgesia (PCA) device with 5 µg/mL fentanyl was used for postoperative analgesia and was administered as a standard procedure to all patients. The bolus dose was set as 10 µg, the louckout time as 5 min, and the one-hour limit as 50 µg. In the event that the Numeric Rating Scale (NRS) pain score ≥ 4, rescue analgesia with IV tramadol 0.5 mg/kg (maximum daily dose 400 mg) was administeredThe total opioid consumption was calculated as morphine milligram equivalents (MME) using the GlobalRPH opioid equivalency calculator. Conversion factors used were:
  * Fentanyl: 0.1 mg IV fentanyl = 10 mg IV morphine
  * Tramadol: 100 mg tramadol = 10 mg morphine

SECONDARY OUTCOMES:
Post-operative acute pain | Postoperative Day 1
  Pain status at rest and while activity (coughing and walking) was assessed by VAS scores at 0, 2, 4, 6, 8, 12 and 24 hours after surgery. The VAS is an 11-point numeric scale which ranges from 0 to 10 at rest and during activity.
The incidences of post-operative nausea and vomiting (PONV) | Postoperative Day 1
  The severity of postoperative nausea and vomiting (PONV) was assessed using a Verbal Descriptive Scale(VDS) at 0, 2, 4, 6, 8, 12 and 24, hours after surgery. If a score of 3 or more is recorded, ondansetron 0,1 mg/kg iv was administered.

CONTACTS AND LOCATIONS:
Overall Officials: ilke tamdoğan, Principal Investigator — ndokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

REFERENCES:
- [Result] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Result] Seyhan TO, Tugrul M, Sungur MO, Kayacan S, Telci L, Pembeci K, Akpir K. Effects of three different dose regimens of magnesium on propofol requirements, haemodynamic variables and postoperative pain relief in gynaecological surgery. Br J Anaesth. 2006 Feb;96(2):247-52. doi: 10.1093/bja/aei291. Epub 2005 Nov 25. PMID 16311277
- [Result] Benevides ML, Fialho DC, Linck D, Oliveira AL, Ramalho DHV, Benevides MM. Intravenous magnesium sulfate for postoperative analgesia after abdominal hysterectomy under spinal anesthesia: a randomized, double-blind trial. Braz J Anesthesiol. 2021 Sep-Oct;71(5):498-504. doi: 10.1016/j.bjane.2021.01.008. Epub 2021 Mar 21. PMID 33762190
- [Result] Sousa AM, Rosado GM, Neto Jde S, Guimaraes GM, Ashmawi HA. Magnesium sulfate improves postoperative analgesia in laparoscopic gynecologic surgeries: a double-blind randomized controlled trial. J Clin Anesth. 2016 Nov;34:379-84. doi: 10.1016/j.jclinane.2016.05.006. Epub 2016 Jun 5. PMID 27687417

DOCUMENTS (3):
  • Study Protocol (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT05644873/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05644873/SAP_001.pdf
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT05644873/ICF_002.pdf